CLINICAL TRIAL: NCT00715936
Title: Phase 1 Study of Integration of Early Child Development Interventions in a Community Health Service in Sindh, Pakistan
Brief Title: The Pakistan Early Childhood Development Scale Up Trial
Acronym: PEDS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: UNICEF (Other)
Responsible Party: Principal Investigator, Dr Aisha Khizar Yousafzai, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 993-PEDS/ERC-08
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Early Child Development and Growth
Keywords: Integrated early child development, growth and health; Psychosocial stimulation; Care for child development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Active Comparator): Routine services for infants and young children delivered by the Lady Health Workers of the National Programme for Family Planning and Primary Healthcare (Basic Health and Nutrition Education and Services)
  Interventions: Behavioral: Control
- ECD Group (Experimental): Stimulation and care for development (plus basic health and nutrition education and services)
  Interventions: Behavioral: ECD
- Enhanced Nutrition (Experimental): Care for Nutrition: Enhanced education messages and Sprinkles for children aged 6-24 months (plus basic health and nutrition education and services)
  Interventions: Behavioral: Enhanced Nutrition
- ECD and Enhanced Nutrition (Experimental): Stimulation and care for development and care for nutrition (plus basic health and nutrition education and services)
  Interventions: Behavioral: ECD; Behavioral: Enhanced Nutrition

INTERVENTIONS:
Behavioral: Control
  Arms: Control
Behavioral: ECD
  Arms: ECD Group; ECD and Enhanced Nutrition
Behavioral: Enhanced Nutrition
  Arms: ECD and Enhanced Nutrition; Enhanced Nutrition

SUMMARY:
The purpose of this study is to evaluate whether the integration of an early child 'stimulation and care for development' intervention, either alone or in combination with an 'enhanced care for nutrition' intervention, delivered by Lady Health Workers to families with infants and young children aged 0-24 months living in rural Sindh in Pakistan, has beneficial outcomes on child development (cognitive, language, motor and social emotional development) and child growth.

DETAILED DESCRIPTION:
In Pakistan, the "National Program for Family Planning and Primary Healthcare" delivers maternal and child health and nutrition services in rural and remote areas of Pakistan through community-based Lady Health Workers. The strengths of the programme include provision of services at grassroots levels, reinforcement of health and basic nutrition messages and community acceptability. Given, the growing recognition that optimal early child development (ECD) also requires the integration of psychosocial care; the PEDS-Trial has been proposed to evaluate the benefits of the addition of 'stimulation and care for development' interventions and the feasibility of scaling up an ECD strategy within the community healthcare system of Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* All children born in the defined geographical area of study during the study enrollment period will be eligible for the study along with their primary care giver (mother). Infant must be 1d-2.5m of age at time of enrolment.

Exclusion Criteria:

* Children born with profound severe disabilities

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1489 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Early Child Development | 24 months of child age
  Cognitive, Language, Motor, Social-Emotional development
Child Growth | 24 months of child age
  Length/Height, Weight, Mid Arm Circumference, Head Circumference

SECONDARY OUTCOMES:
Caregiving Mediators: Maternal Psychological Distress (Depression) | Baseline, 6 months, 12 months, 18 months and 24 months of child age
  Self-Reporting Questionnaire (SRQ)-20
Caregiving mediators: Caregiving Environment | 6 months and 18 months of child age
  Home Observation and Measurement of the Environment (HOME) Inventory
Caregiving Mediator: Mother/Child Interaction | 12 months and 24 months of child age
  Live observation
Caregiving Mediator: Care for Development | Baseline, 12 months and 24 months of child age
  Knowledge and Practices Questionnaire (Maternal Report)
Caregiving Mediator: Feeding Practices | Baseline, 6 months, 12 months, 18 months and 24 months of child age
  Maternal report of infant and young child feeding practices
Morbidity | Monthly report
  Maternal recall
Anaemia Status | 24 months child age
  Haemoglobin assessment using HemoCue Assay

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, MBBS, PhD, Study Chair — Aga Khan University; Aisha K Yousafzai, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Project Office, Dept of Paediatrics and Child Health, AKU, Naushero Feroze, Sindh, Pakistan

REFERENCES:
- [Derived] Yousafzai AK, Obradovic J, Rasheed MA, Rizvi A, Portilla XA, Tirado-Strayer N, Siyal S, Memon U. Effects of responsive stimulation and nutrition interventions on children's development and growth at age 4 years in a disadvantaged population in Pakistan: a longitudinal follow-up of a cluster-randomised factorial effectiveness trial. Lancet Glob Health. 2016 Aug;4(8):e548-58. doi: 10.1016/S2214-109X(16)30100-0. Epub 2016 Jun 21. PMID 27342433
- [Derived] Yousafzai AK, Rasheed MA, Rizvi A, Armstrong R, Bhutta ZA. Effect of integrated responsive stimulation and nutrition interventions in the Lady Health Worker programme in Pakistan on child development, growth, and health outcomes: a cluster-randomised factorial effectiveness trial. Lancet. 2014 Oct 4;384(9950):1282-93. doi: 10.1016/S0140-6736(14)60455-4. Epub 2014 Jun 16. PMID 24947106